CLINICAL TRIAL: NCT03302403
Title: Clinical Study of Redirected Autologous T Cells With a Chimeric Antigen Receptor in Patients With Malignant Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kang YU (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kang YU, Head of Department of Hematology, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGZ001
Record Dates: First submitted 2017-09-26; First posted 2017-10-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: B Cell Lymphoma; B Cell Leukemia; Myeloma; Hepatocellular Carcinoma; Pancreatic Carcinoma; Adenocarcinoma of Esophagogastric Junction
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Neoplasms, Plasma Cell; Carcinoma, Hepatocellular; Pancreatic Neoplasms | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T cell (Experimental): In this study, autologous T cells transduced with a chimeric antigen receptor are used to treat patients with malignant tumors:
  CAR-CD19 T cell is for the treatment of B-cell Leukaemia/Lymphoma; CAR-BCMA T cell is for the treatment of Myeloma; CAR-GPC3 T cell is for the treatment of Hepatocellular Carcinoma; CAR-CLD18 T cell is for the treatment of Pancreatic Carcinoma and Adenocarcinoma of Esophagogastric Junction.
  Route of administration: Intravenous injection.
  Lymphodepletion conditioning:
  Lymphodepletion will be conducted several days prior to CAR T cell infusion, which may improve in vivo cell count and survival of T cells.
  A combination of fludarabine and cyclophosphamide will be used for lymphodepletion.
  Interventions: Genetic: CAR-CD19 T cell; Genetic: CAR-BCMA T cell; Genetic: CAR-GPC3 T cell; Genetic: CAR-CLD18 T cell; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: CAR-CD19 T cell — Self-controlled dose escalation and classic "3+3" dose escalation will be applied.
  Other Names: CD19-redirected Autologous Cell
Genetic: CAR-BCMA T cell — Self-controlled dose escalation and classic "3+3" dose escalation will be applied.
  Other Names: BCMA-redirected Autologous Cell
Genetic: CAR-GPC3 T cell — Self-controlled dose escalation and classic "3+3" dose escalation will be applied.
  Other Names: GPC3-redirected Autologous Cell
Genetic: CAR-CLD18 T cell — Self-controlled dose escalation and classic "3+3" dose escalation will be applied.
  Other Names: Claudin18.2-redirected Autologous Cell
Drug: Fludarabine — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety, efficacy and cytokinetics of CAR T cells in patients with malignant tumors with positive antigen targets.

CAR T cells are genetically engineered to express single-chain variable fragment (scFv) targeting indication-specific antigens.

The investigational CAR T cells and proposed indications are as follows:

CAR-CD19 T cells for B cell leukaemia/lymphoma; CAR-BCMA T cells for myeloma; CAR-GPC3 T cell for hepatocellular carcinoma; CAR-CLD18 T cells for pancreatic carcinoma and adenocarcinoma of esophagogastric junction.

DETAILED DESCRIPTION:
This study is designed to determine the safety, tolerability and engraftment potential of lentivirus-transduced CAR T cells in patients with malignant tumors.

Primary objectives:

1. Determine the safety and tolerability of CAR T cells (autologous T cells transduced with chimeric antigen receptors recognizing CD19, BCMA, GPC3 and Claudin18.2) in patients with malignant tumors (B-cell lymphoblastic leukaemia/lymphoma, myeloma, hepatocellular carcinoma, pancreatic carcinoma and adenocarcinoma of esophagogastric junction).
2. Observe the cytokinetics of CAR T cells.

Secondary objectives:

1. Observe the efficacy of CAR T cells in patients with malignant tumors.
2. Make an evaluation on the distribution and in vivo survival of CAR T cells in targeted tissues.
3. Observe the immunogenicity of CAR T cells, and determine if there are anti-scFv cellular immune response and anti-scFv humoral immune response.
4. Observe the changes of cell subsets for CAR T cells against T cells (Tcm, central memory T lymphocytes; Tem, effector memory T lymphocytes; Treg, regulatory T-lymphocytes).

ELIGIBILITY:
Inclusion Criteria:

I. B-Cell Lymphoblastic Leukaemia/Lymphoma

1. Patients aged between 18 ~ 65 with B-cell lymphoblastic leukaemia/lymphoma.
2. CD19-positive B-cell lymphoblastic leukaemia/lymphoma.
3. Patients with unmet medical needs for which there are no effective therapies known at this time:

   A. Relapsed or Refractory (r/r) Acute Lymphoblastic Leukemia (ALL)

   Patients with r/r ALL for whom hematopoietic stem cell transplantation (HSCT) is not suitable due to following reasons:
   1. Age;
   2. Excessive tumor burden or concomitant disease;
   3. No donor available.

   B. CD19-positive Follicular Lymphoma:
   1. At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy;
   2. Less than 6 months between last chemotherapy and disease progression (most recent progression free interval < 6 months);
   3. Disease progression after most recent systemic therapy (chemotherapy, MoAb, etc.).

   C. Chronic Lymphocytic Leukemia (CLL)
   1. At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy);
   2. Less than6 months between last chemotherapy and disease progression (most recent progression free interval < 6 months);
   3. Not eligible or appropriate for conventional HSCT.
   4. Disease progression after most recent systemic therapy (chemotherapy, MoAb, etc.).

   D. Mantle Cell Lymphoma
   1. At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy);
   2. Disease progression after most recent systemic therapy (chemotherapy, MoAb, etc.)；
   3. Relapsed after prior autologous SCT.

   E. B-Cell Prolymphocytic Leukemia (PLL)

   Relapsed or residual disease after at least 1 prior therapy and not eligible for HSCT.

   F. CD19-positive Diffuse Large B Cell Lymphoma
   1. At least 2 prior chemotherapy regimens (not including single agent monoclonal antibody (Rituxan) therapy;
   2. Stage III-IV disease.
   3. Less than 6 months between last chemotherapy and disease progression (most recent progression free interval < 6 months);
   4. Disease progression after most recent therapy (chemotherapy, MoAb, etc.).
4. Expected survival > 12 weeks.
5. At least one measurable lesion (≥ 10 mm) for patients with lymphoma.
6. ECOG scores 0-1, or KPS scores > 70.
7. Adequate venous access for apheresis or venous sampling, and no other contraindications for leukapheresis.
8. WBC ≥ 2.5×10^9/L; PLT ≥ 60×10^9/L (for patients with lymphoma); Hb ≥ 9.0 g/dL; LY ≥ 0.47×10^9/L; LY% ≥ 15%.
9. Serum Alb ≥ 30 g/L.
10. Serum creatinine ≤ 1.5 ULN.
11. ALT ≤ 2.5 ULN; AST ≤ 2.5 ULN.
12. Serum total bilirubin ≤ 1.5 ULN. The above lab results should not include those obtained from continuous supportive treatment that is ongoing.

II. Myeloma

1. Patients aged between 18 ~ 75 with relapsed or refractory multiple myeloma.
2. Bone marrow sample is confirmed as BCMA-positive by flow cytometry or pathological examination.
3. Patients with relapsed or refractory malignancies who meet the following descriptions:

   1. Curative efficacy is little or disease progressed after 2 courses of standard treatment regimen;
   2. Disease relapsed after chemotherapy or HSCT. Curative efficacy is little or disease progressed after 2 courses of original treatment regimen;
   3. More than 30 days between last treatment and disease progression;
   4. There is no indication for HSCT at present;
   5. Disease progression is defined as per "Chinese Guidelines for Diagnosis and Treatment of Multiple Myeloma (Version 2015)". One or more of the following conditions should be met:

   i. Serum M-protein increases ≥ 25% (absolute increase should be ≥ 5 g/L). If serum M protein is ≥ 50 g/L at baseline, increase of serum M protein can be ≥ 10 g/L; ii. Urine M-protein increases ≥ 25% (absolute increase should be ≥ 200 mg/24 h); iii. If the serum and urine M-protein are not detectable, a ≥ 25% increase in the difference between involved and uninvolved FLC levels is required (absolute increase should be ≥ 100 mg/L); iv. Bone marrow plasma cell percentage increases ≥ 25% (absolute increase should be ≥ 10%); v. Size of existing bone lesions or soft tissue plasmacytomas increased by ≥ 25%, or development of new lytic bone lesions or oft tissue plasmacytomas; vi. Development of hypercalcemia that can be attributed to plasma cell proliferative disorder (corrected calcium is > 2.8 mmol/L or 11.5 mg/dL).
4. Expected survival > 12 weeks.
5. Disease is measurable, and at least one of the following conditions should be satisfied:

   1. Serum M-protein is ≥ 10 g/L;
   2. 24-hour urine M-protein is ≥ 200 mg;
   3. Serum FLC is ≥ 5 mg/dL;
   4. Plasmacytomas that can be measured or evaluated by imaging;
   5. Bone marrow plasma cell percentage is ≥ 20%.
6. ECOG scores 0 - 1 or CCI scores ≤ 2.
7. Adequate venous access for apheresis and venous blood sampling, and no other contraindications for leukapheresis.
8. WBC ≥ 1.5×10^9/L; PLT ≥ 45×10^9/L; Hb ≥ 9.0 g/dL.
9. Serum creatinine ≤ 1.5 ULN.
10. ALT ≤ 2.5 ULN; AST ≤ 2.5 ULN. The above lab results should not include those obtained from continuous supportive treatment that is ongoing.

III. Hepatocellular Carcinoma (HCC)

1. Patients aged 18 ~ 70 with refractory hepatocellular carcinoma.
2. Patients with HCC that cannot be eradicated by resection who have received ablation or resection in the last 4 to 12 weeks.
3. IHC testing confirmed as GPC3-positive HCC.
4. Expected survival > 12 weeks.
5. At least one measurable lesion (≥ 10 mm).
6. Cirrhosis of the liver: Child-Pugh Class A, or Child-Pugh Class B scored at 7.
7. ECOG scores 0 - 1 or KPS scores > 70.
8. Adequate venous access for apheresis and venous blood sampling, and no other contraindications for leukapheresis.
9. Hematology:

   WBC ≥ 2.5×10^9/L; PLT ≥ 60×10^9/L; Hb ≥ 9.0 g/dL; MID ≥ 1.0×10^9/L; LY ≥ 0.4×10^9/L.
10. Blood Chemistry:

    Serum Alb ≥ 30 g/L; Serum lipase and serum amylase < 1.5 ULN; Serum creatinine ≤ 1.5 ULN; ALT ≤ 5 ULN; AST ≤ 5 ULN; Serum total bilirubin ≤ 2.5 ULN.
11. Coagulation Test:

    Prothrombin time is at most 4 seconds longer than normal value.
12. Able to understand and sign the informed consent. All test results should be within their normal ranges, and patients are not receiving continuous supportive treatment.

IV. Pancreatic Carcinoma and Adenocarcinoma of Esophagogastric Junction

1. Patients aged 18 ~ 70 with pathologically confirmed advanced pancreatic carcinoma and adenocarcinoma of esophagogastric junction.
2. IHC testing confirmed as Claudin18.2 positive.
3. Patients with advanced pancreatic carcinoma and adenocarcinoma of esophagogastric junction that cannot be eradicated by resection.
4. Expected survival after first dose of study drug > 12 weeks.
5. At least one measurable lesion (≥ 10 mm) available for imaging assessment.
6. ECOG scores 0 - 1.
7. Adequate venous access for apheresis and venous blood sampling, and no other contraindications for leukapheresis.
8. WBC ≥ 2.5×10^9/L; PLT ≥ 100×10^9/L; Hb ≥ 9.0 g/dL; MID ≥ 1.5×10^9/L; LY ≥ 0.47×10^9/L; LY% ≥ 15%.
9. Serum Alb ≥ 30 g/L.
10. Serum lipase and serum amylase < 1.5 ULN.
11. Serum creatinine ≤ 1.5 ULN.
12. ALT ≤ 2.5 ULN; AST ≤ 2.5 ULN; If osseous metastasis or liver metastasis is developed and alkaline phosphatase is > 2.5 ULN, than ALT and AST should be < 1.5 ULN.
13. Serum total bilirubin ≤ 1.5 ULN.
14. PT: INR < 1.7; PT < (ULN + 4) s All test results should be within their normal ranges, and patients are not receiving continuous supportive treatment.

Exclusion Criteria:

Patients with any of the following conditions are not eligible for this study.

1. Transduction of target lymphocytes < 10%, expansion in response to αCD3/CD28 costimulation < 5-fold.
2. Pregnant or lactating women.
3. HIV positive, or HCV positive
4. Uncontrolled active infection, including active tuberculosis and HBV DNA copies ≥ 1×10^3 copies/mL.
5. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
6. Allergic to immunotherapies and related drugs.
7. Patients with heart disease for which treatment is needed or with poorly controlled hypertension.
8. Hyponatremia: serum sodium level < 125 mmol/L.
9. Baseline serum potassium < 3.5 mmol/L (taking potassium supplements before participating in the study to raise potassium level is acceptable).
10. Previous treatment with chemoradiotherapy, immunotherapy and tumor-targeting drug conducted 2 weeks prior to participation in this study or blood collection.
11. Patients have undertaken immunosuppressor for graft-versus-host disease (GVHD) within 4 weeks before participation in this study or blood collection, or the patient is diagnosed with acute or chronic GVHD.
12. Other severe disease that may restrain patients from participating in this study (e.g. diabetes, severe cardiac dysfunction, myocardial infarction or unstable arrhythmias or unstable angina in recent 6 months, gastric ulcer, active autoimmune disease, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2020-12-12 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with CRA T-related adverse events as assessed by CTCAE v4.03 | 24 weeks
  Number of participants with study related adverse events which are defined as laboratory toxicities and clinical events that are possible, likely or definitely related to study treatment at any time from the infusion until week 24, including infusion related toxicity and any toxicity possibly related to CAR T cells.

SECONDARY OUTCOMES:
Engraftment | 2 years
  Duration of in vivo survival of CAR T cells is defined as "engraftment". The primary engraftment endpoint is the number of DNA vector copies per mL blood of CAR T cells at regular intervals through 24 hours following the initial infusion. PCR for CAR T vector sequences will be performed until any 2 sequential tests are negative, documented as engraftment of CAR T cells.

OTHER OUTCOMES:
Progression-free Survival (PFS) | 5 years for BCMA, 2 years for GPC3, CD19 and Claudin 18.2
  Determine anti-tumor responses to CAR T cell infusion by the length of time during and after the treatment of the malignancy that the patient lives with the disease but it does not get worse.
Time to Tumor Progression (TTP) | 5 years for BCMA, 2 years for GPC3, CD19 and Claudin 18.2
  Determine anti-tumor responses to CAR T cell infusion by time to tumor progression.
Disease Control Rate (DCR) | 2 years
  Determine anti-tumor responses to CAR T cell infusion by proportion of patients who demonstrate response to treatment.
Objective Remission Rate (ORR) | 2 years
  Determine anti-tumor responses to CAR T cell infusion by percentage of patients who have achieved complete response or partial response.
Overall survival (OS) | 5 years for BCMA, 2 years for GPC3, CD19 and Claudin 18.2
  Determine anti-tumor responses to CAR T cell infusion by time from study enrollment until death.
Number of DNA copies of CAR T cells in tissue samples | 2 years
  The number of DNA copies of CAR-BCMA T cells in lymph node samples or bone marrow samples at regular intervals through 24 hours following the initial infusion.
Anti-drug antibody | 2 years
  Detect positive rate and titer of anti-drug antibody (ADA).
Changes of cell subsets for CAR T cells against T cells | 2 years
  Observe the changes of cell subsets for CAR T cells against T cells (Tcm, central memory T lymphocytes; Tem, effector memory T lymphocytes; Treg, regulatory T-lymphocytes).

CONTACTS AND LOCATIONS:
Overall Officials: Mengtao Zhou, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Kang Yu, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University; Songfu Jiang, MD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dong R, Jiang S, Chen Y, Ma Y, Sun L, Xing C, Zhang S, Yu K. Prognostic Significance of Cytokine Release Syndrome in B Cell Hematological Malignancies Patients After Chimeric Antigen Receptor T Cell Therapy. J Interferon Cytokine Res. 2021 Dec;41(12):469-476. doi: 10.1089/jir.2021.0057. PMID 34935483